CLINICAL TRIAL: NCT05786547
Title: Varenicline and Mobile Behavioral Assistance for Tobacco Cessation in HIV Care in India
Brief Title: V+PSF-M for Tobacco Cessation in HIV Care in India
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-1017; 1U01CA261614-01 (NIH)
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Human Immunodeficiency Virus; Smoking Cessation; Smoking, Tobacco
Keywords: Human Immunodeficiency Virus; Smoking Cessation; Smoking, Tobacco
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Smoking Cessation; Tobacco Smoking | interventions — Varenicline; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varenicline + Positively Smoke Free - Mobile (Experimental): Offer of varenicline per package dosing with dose escalation over week 1: 0.5 mg once daily on days 1 - 3, 0.5 mg twice daily on days 4 -7, followed by 1.0 mg twice daily on days 8 to 84.
  Offer of Positively Smoke Free Mobile delivered by mobile phone including 42 days of content, tailored to individual quit date.
  Interventions: Drug: Varenicline; Behavioral: Positively Smoke Free Mobile (PSF-M)
- Standard Care (Active Comparator): Brief advice to quit tobacco Offer of referral to the national tobacco quitline
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Drug: Varenicline — Per package dosing, tablet taken orally
  Other Names: Champix, apovarenicline, Nocrav
  Arms: Varenicline + Positively Smoke Free - Mobile
Behavioral: Positively Smoke Free Mobile (PSF-M) — Behavioral tobacco cessation intervention for people living with HIV, delivered via mobile phone
  Arms: Varenicline + Positively Smoke Free - Mobile
Behavioral: Standard Care — Brief cessation advice plus referral to local tobacco quitline
  Arms: Standard Care

SUMMARY:
The goal of this research study is to test an intervention to help quit tobacco use in participants with Human Immunodeficiency Virus (HIV).

The study interventions used in this research study are:

* Positively Smoke Free - Mobile (PSF-M) (mobile behavioral program)
* Varenicline (or Chantix, apovarenicline, Champix or Nocrav)

DETAILED DESCRIPTION:
Open-label, practice-based randomized trial of varenicline + Positively Smoke Free-Mobile (PSF-M) for people living with Human Immunodeficiency Virus (PWH) who smoke or use both smoked and smokeless tobacco compared with a group that receives standard care including brief advice and quitline referral.

Positively Smoke Free (PSF) is a behavioral intervention which has been tested in multiple formats including a mobile version. Varenicline is the single most-effective pharmacotherapy agent for quitting tobacco with demonstrated efficacy for cessation of cigarettes, smokeless tobacco, and cessation among smokers with comorbidities

In this study, participants will be randomized to either Group 1: Varenicline + Positively Smoke Free-Mobile adapted for Chennai versus Group 2: Standard care with brief tobacco cessation advice and referral to the national quitline.

Research procedures include screening for eligibility, in-clinic visits, and completion of surveys and questionnaires.

Participation in this study is expected to last about 24 weeks.

It is expected about 400 people will take part in this research study.

This study is funded by the National Cancer Institute of the National Institute of Health (NIH).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Confirmed HIV diagnosis
* Self-reported current smoking or dual tobacco use verified either by exhaled carbon monoxide ≥7 ppm, or by positive qualitative cotinine point-of-care test
* Able to read at 6th grade level or greater and speak Tamil, Telugu or English
* Able to use varenicline safely based on evaluation by primary provider at VHS
* Women of childbearing potential who consent to use a medically approved method of contraception or abstain from intercourse while taking study medication and for one month after.
* Ready to quit or interested in quitting

Exclusion Criteria:

* Pregnant or planning to become pregnant in the next 6 months
* Breastfeeding
* Myocardial infarction in past 30 days or unstable angina
* History of liver or kidney failure
* Alanine aminotransferase and Aspartate aminotransferase > 2 times upper limit of normal or creatinine clearance <50 in past 6 months
* History of suicide attempt
* Current suicidal ideation
* Untreated or unstable major depressive disorder
* History of psychosis or on anti-psychotic medications
* Cognitive impairment limiting ability to consent
* Allergy to varenicline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
7-Day Point Prevalent Abstinence Rate | 24 weeks post-randomization
  Defined as abstinence from all combustible and smokeless tobacco products in the 7 days preceding 24-week follow-up supported by a negative urine cotinine test of < 50 ng/ml

SECONDARY OUTCOMES:
7-day self-reported Point Prevalent Abstinence Rate | 4 weeks post-randomization
  Defined as abstinence from all combustible and smokeless tobacco products in the 7 days preceding follow-up
7-day self-reported Point Prevalent Abstinence Rate | 12 weeks post-randomization
  Defined as abstinence from all combustible and smokeless tobacco products in the 7 days preceding 24-week follow-up supported by a negative urine cotinine test of < 50 ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Gina Kruse, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- University of Colorado, Aurora, Colorado, United States
- VHS Infectious Disease Medical Centre, CART Clinical Research Site, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Principle Investigator. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation.

REFERENCES:
- [Derived] Malpeddi T, Poongulali S, Shuter J, Rigotti NA, An LC, Kumarasamy N, Reddy KP, Shergina E, Colborn K, Faith B, Sierra YL, Kruse GR. Protocol for the Mobile behavioral support plus varenicline for tobacco cessation among people living with HIV in India (MoVIe): A hybrid implementation-effectiveness randomized trial. Contemp Clin Trials. 2026 Jan;160:108179. doi: 10.1016/j.cct.2025.108179. Epub 2025 Dec 4. PMID 41352530